CLINICAL TRIAL: NCT02441621
Title: Prediction of Fluid Responsiveness in Presence of Diastolic Dysfunction
Brief Title: Prediction of Volume Responsiveness in Presence of Left Ventricular Diastolic Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Ole Broch, MD, MD, University Hospital Schleswig-Holstein
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AZ-139
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Hemodynamics
Keywords: fluid responsiveness; diastolic dysfunction; left ventricular
MeSH Terms: interventions — Premedication; Intubation; Respiration, Artificial; Central Venous Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Passive leg raising (Other)
  Interventions: Other: passive leg raising
- premedication (Other)
  Interventions: Other: premedication
- intubation and mechanical ventilation (Other)
  Interventions: Other: intubation and mechanical ventilation
- central venous catheter (Other)
  Interventions: Other: central venous catheter
- arterial catheter (Other): Continuous monitoring is performed including electrocardiogram, radial arterial pressure catheter
  Interventions: Other: arterial catheter
- transesophageal echocardiography (Other)
  Interventions: Other: transesophageal echocardiography
- transpulmonary thermodilution catheter (Other)
  Interventions: Other: transpulmonary thermodilution catheter

INTERVENTIONS:
Other: passive leg raising — The passive leg raising maneuver (PLR) involves a leg elevation up to 45° with the trunk in a horizontal position and is performed to induce hemodynamic effects by a volume challenge, turning unstressed blood volume to stressed volume proportional to body size.
  Arms: Passive leg raising
Other: premedication — patients receive premedication with midazolam 7.5 mg p.o.
  Arms: premedication
Other: intubation and mechanical ventilation — After induction of anesthesia with sufentanil (0.5 µg/kg) and propofol (1.5 mg/kg), orotracheal intubation is facilitated with rocuronium (0.6 mg/kg). Anesthesia is maintained with sufentanil (1 µg/kg/h) and propofol (3 mg/kg/h) and patients are ventilated with an oxygen/air mixture in volume-controlled mode, using a tidal volume of 8 ml/kg related to the ideal body weight. Positive end-expiratory pressure is set at 5 cmH2O.
  Arms: intubation and mechanical ventilation
Other: central venous catheter — a central venous catheter in the right or left internal jugular vein.
  Arms: central venous catheter
Other: arterial catheter — Continuous monitoring is performed including electrocardiogram, radial arterial pressure catheter
  Arms: arterial catheter
Other: transesophageal echocardiography — Before placement of a transpulmonary thermodilution catheter a transesophageal echocardiography (TOE) is performed. TOE is used to detect diastolic dysfunction of the left ventricle and to exclude right ventricular dysfunction.
  Arms: transesophageal echocardiography
Other: transpulmonary thermodilution catheter — In presence of left ventricular dysfunction a transpulmonary thermodilution catheter is placed in the femoral artery and connected to a PiCCO2 monitor (PiCCO2, Pulsion Medical Systems, Munich, Germany).
  Arms: transpulmonary thermodilution catheter

SUMMARY:
The ability of the global end-diastolic volume index (GEDVI), stroke volume variation (SVV) and pulse pressure variation (PPV) for prediction of fluid responsiveness in presence of left ventricular diastolic dysfunction is still unknown. The aim of the present study was to challenge the predictive power of GEDVI, SVV and PPV in cardiac surgery patients undergoing aortic valve replacement.

DETAILED DESCRIPTION:
All patients receive premedication with midazolam 7.5 mg p.o.. After induction of anesthesia with sufentanil (0.5 µg/kg) and propofol (1.5 mg/kg), orotracheal intubation is facilitated with rocuronium (0.6 mg/kg). Anesthesia is maintained with sufentanil (1 µg/kg/h) and propofol (3 mg/kg/h) and patients are ventilated with an oxygen/air mixture in volume-controlled mode, using a tidal volume of 8 ml/kg related to the ideal body weight. Positive end-expiratory pressure is set at 5 cmH2O. Continuous monitoring is performed including electrocardiogram, radial arterial pressure catheter and a central venous catheter in the right or left internal jugular vein. Before placement of a transpulmonary thermodilution catheter a transesophageal echocardiography (TOE) is performed. TOE is used to detect diastolic dysfunction of the left ventricle and to exclude right ventricular dysfunction. In presence of left ventricular dysfunction a transpulmonary thermodilution catheter is placed in the femoral artery and connected to a PiCCO2 monitor (PiCCO2, Pulsion Medical Systems, Munich, Germany). Additionally capnography, urine output, temperature (blood, bladder and nasopharyngeal), airway pressure, and pulse oximetry are recorded.

Before starting operation a passive leg raising is performed. The passive leg raising maneuver (PLR) involves a leg elevation up to 45° with the trunk in a horizontal position and was performed to induce hemodynamic effects by a volume challenge, turning unstressed blood volume to stressed volume proportional to body size. In case of an increase of stroke volume index (SVI) >15% during PLR, patients were defined as responders.

All patients were studied with no changes in anesthesia management. Measurements of SVI, GEDVI, SVV and PPV are performed before, during and after PLR. Thereafter, patients receive a fluid Bolus of 500 ml crystalloids. Again, measurements are performed before and after fluid replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 yrs of age
* Patients with a left ventricular ejection fraction ≥0.5
* Patients with left ventricular diastolic dysfunction.

Exclusion Criteria:

* Emergency procedures
* Right ventricular dysfunction
* Hemodynamic instability requiring pharmacologic Support
* Ongoing arrhythmia
* Intracardiac Shunts
* Severe mitral stenosis or insufficiency
* Aortic aneurysm > 4 cm
* Use of an artificial left ventricular assist device or intra - aortic balloon pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Increase in stroke volume index (SVI) >15% | Patients will be obtained until the end of the operation, an expected average of 5 hours
  In presence of an increase of SVI >15% during PLR and/or 500 ml crystalloids, patients are defined as responders.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Broch, MD, Principal Investigator — Consultant anesthetist
Locations (1):
- Ole Broch, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Rex S, Schalte G, Schroth S, de Waal EE, Metzelder S, Overbeck Y, Rossaint R, Buhre W. Limitations of arterial pulse pressure variation and left ventricular stroke volume variation in estimating cardiac pre-load during open heart surgery. Acta Anaesthesiol Scand. 2007 Oct;51(9):1258-67. doi: 10.1111/j.1399-6576.2007.01423.x. Epub 2007 Aug 20. PMID 17714575
- [Background] Hofer CK, Muller SM, Furrer L, Klaghofer R, Genoni M, Zollinger A. Stroke volume and pulse pressure variation for prediction of fluid responsiveness in patients undergoing off-pump coronary artery bypass grafting. Chest. 2005 Aug;128(2):848-54. doi: 10.1378/chest.128.2.848. PMID 16100177
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Renner J, Gruenewald M, Brand P, Steinfath M, Scholz J, Lutter G, Bein B. Global end-diastolic volume as a variable of fluid responsiveness during acute changing loading conditions. J Cardiothorac Vasc Anesth. 2007 Oct;21(5):650-4. doi: 10.1053/j.jvca.2007.05.006. Epub 2007 Jul 16. PMID 17905268
- [Background] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963
- [Background] Osman D, Ridel C, Ray P, Monnet X, Anguel N, Richard C, Teboul JL. Cardiac filling pressures are not appropriate to predict hemodynamic response to volume challenge. Crit Care Med. 2007 Jan;35(1):64-8. doi: 10.1097/01.CCM.0000249851.94101.4F. PMID 17080001
- [Background] Mahjoub Y, Pila C, Friggeri A, Zogheib E, Lobjoie E, Tinturier F, Galy C, Slama M, Dupont H. Assessing fluid responsiveness in critically ill patients: False-positive pulse pressure variation is detected by Doppler echocardiographic evaluation of the right ventricle. Crit Care Med. 2009 Sep;37(9):2570-5. doi: 10.1097/CCM.0b013e3181a380a3. PMID 19623051
- [Background] Cioffi G, Mazzone C, Barbati G, Rossi A, Nistri S, Ognibeni F, Tarantini L, Di Lenarda A, Faggiano P, Pulignano G, Stefenelli C, de Simone G, Devereux RB. Combined circumferential and longitudinal left ventricular systolic dysfunction in patients with asymptomatic aortic stenosis. Echocardiography. 2015 Jul;32(7):1064-72. doi: 10.1111/echo.12825. Epub 2014 Nov 5. PMID 25370995
- [Background] Rader F, Sachdev E, Arsanjani R, Siegel RJ. Left ventricular hypertrophy in valvular aortic stenosis: mechanisms and clinical implications. Am J Med. 2015 Apr;128(4):344-52. doi: 10.1016/j.amjmed.2014.10.054. Epub 2014 Nov 25. PMID 25460869